CLINICAL TRIAL: NCT06227949
Title: FSH and LH Versus FSH Alone for Ovarian Stimulation in Non-hormone Sensitive Onco-fertility Patients: an Exploratory Randomized Controlled Trial
Brief Title: FSH and LH Versus FSH Alone for Ovarian Stimulation in Non-hormone Sensitive Onco-fertility Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ellen Greenblatt (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor-Investigator, Ellen Greenblatt, Professor, Mount Sinai Hospital, Canada
Organization: Mount Sinai Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200061_0066
Record Dates: First submitted 2023-12-21; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Fertility Preservation
Keywords: IVF; fertility preservation; oncofertility; rLH; FSH; cryopreservation
MeSH Terms: interventions — Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned in a 1:1 ratio to either treatment or control group. Treatments in each of the trial arms will be as follows:
  1. Treatment arm: Patients will self-administer a subcutaneous injection of Gonal-F (FSH) in addition to Luveris daily until a pre-set criteria to trigger ovulation is reached.
  2. Control arm: Patients will self-administer a subcutaneous injection of Gonal-F (FSH) daily until a pre-set criteria to trigger ovulation is reached.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): subcutaneous injection of Gonal-F (FSH)
- Intervention (Experimental): subcutaneous injection of Luveris in addition to Gonal-F (FSH)
  Interventions: Drug: Luveris

INTERVENTIONS:
Drug: Luveris — Patients will self-administer a subcutaneous injection of Luveris in addition to Gonal-F (FSH) daily until a pre-set criteria to trigger ovulation is reached.
  Arms: Intervention

SUMMARY:
Fertility preservation has been performed before the initiation of cancer therapy as cancer therapy is known to be toxic for ovarian function. However, recent studies have shown that ovarian function is reduced in cancer patients even before they start cancer therapy. Reduced ovarian function has been shown by these patients having fewer mature oocytes (female eggs) and lower peak levels of estradiol (a type of estrogen hormone important for fertility). Other studies have shown that in some types of cancers, cancer patients have lower levels of anti-Müllerian hormone, which is a hormone measured to assess how many eggs patient has remaining in the body. Because of these poorer fertility markers shown in cancer patients prior to therapy, some doctors and researchers believe that alternative medications for stimulating ovaries may prove to be beneficial for stimulating the ovaries during fertility preservation.

Currently, luteinizing hormone injections are approved by Health Canada for patients with hypothalamic dysfunction. Hypothalamic dysfunction is a condition whereby lower levels of fertility hormones are produced because of brain dysfunction. Other reasons luteinizing hormone is used in clinical practice is in patients with poor ovarian reserve and patients who are older.

Recent research studies have suggested that some oncology patients may be poor responders prior to cancer therapy because of their underlying disease. The exact reasons for this poor response are not known. However, some researchers believe it may be related to the interactions between the brain and fertility organs, similar to patients with hypothalamic dysfunction. Because of this possible similarity to patients with hypothalamic dysfunction, adding luteinizing hormone to follicle-stimulating hormone (the hormone typically used for ovarian stimulation) may be beneficial for fertility preservation. Studies have also shown improved fertility outcomes with the addition of luteinizing hormone in non-cancer patients who were previously known to be poor responders to ovarian stimulation.

The clinical trial team is aiming to conduct a randomized controlled trial to evaluate the safety and efficacy of luteinizing hormone in non-hormone sensitive cancer patients (patients with cancer other than the breast, ovary or uterus).

DETAILED DESCRIPTION:
The proposed study is a superiority, randomized controlled trial examining the effect of FSH and rLH (Luveris) versus FSH alone on the number of mature oocytes available for cryopreservation in non-hormone sensitive onco-fertility patients. These patients include those diagnosed with malignancy other than breast, uterine and ovarian cancer.

Given that the care of oncology patients is time sensitive, a random start of the treatment cycle is the usual approach in Mount Sinai Fertility clinic, with no prior priming. The patient has a random serum levels of estrogen, progesterone, LH, FSH and HCG levels. A transvaginal ultrasound is performed as well, and the stage of the cycle is determined. Based on the stage of the cycle, gonadotropin starting time is planned accordingly.

* Early follicular phase: Gonadotropin stimulation started. A GnRH antagonist will be given once the dominant follicle measures >1.4 cm.
* Mid to late follicular phase: patients who have a dominant follicle >1.5 cm with an E2 >300 and a progesterone <5 will be triggered usually with HCG (Ovidrel 250 mcg subcutaneous). After three days gonadotropin stimulation is started.
* Start of luteal phase: start gonadotropin stimulation and once the dominant follicle measure >1.4, a GnRH antagonist will be given.

Patients will be randomly assigned in a 1:1 ratio to either treatment or control group. Treatments in each of the trial arms will be as follows:

1. Treatment arm: Patients will self-administer a subcutaneous injection of Gonal-F (FSH) in addition to Luveris daily until a pre-set criteria to trigger ovulation is reached.
2. Control arm: Patients will self-administer a subcutaneous injection of Gonal-F (FSH) daily until a pre-set criteria to trigger ovulation is reached.

Transvaginal ultrasound and bloodwork monitoring is initiated to monitor the ovarian response.

Once the patient meets one of the following two criteria

1. A serum estradiol (E2) of greater than 2,000 pmol/L
2. A follicle measuring greater than 14 mm,

A daily, subcutaneous injection of a GnRH antagonist (Cetrotide or Ganirelix 0.25 mg) will be administered by the patient subcutaneously to prevent an endogenous surge in LH. Monitoring of the ovarian response will continue until there are 3 or more follicles visualized by transvaginal ultrasound with a mean diameter of ≥17 mm. Ovulation will be subsequently triggered with a subcutaneous injection of HCG or GnRH agonist depending on the managing IVF physician. Twelve hours after their trigger medication, patients will return to the clinic for standard blood work including LH and progesterone. This is a standard confirmatory blood test to confirm that an endogenous LH surge has occurred. In approximately less than 5% of cases, the GnRH-a trigger fails to elicit an optimal surge, which may require a "rescue" low-dose hCG trigger to be administered 24 hours following the initial trigger. The decision to administer a "rescue" trigger will be at the discretion of the managing IVF physician. Transvaginal, ultrasound-guided oocyte retrieval will be performed approximately 36 hours following the administration of the initial trigger.

Once the oocytes are retrieved, the availability of sperm will determine whether the partner's sperm or donor sperm will be used. If the patient desires to cryopreserve oocytes, mature oocytes will be cryopreserved by vitrification process. If embryo cryopreservation is planned, the retrieved oocytes will be fertilized in the lab using traditional IVF or ICSI. Embryos will be grown to day 5 and all "good quality" blastocysts will be cryopreserved using vitrification. At Mount Sinai Fertility clinic, day 5/6 embryos are considered "good quality" for cryopreservation if they are at least a grade 2BB (or above) on day 5 and/or a 3CC (or above) on day 6, according to the classification system by Gardner and Schoolcraft, 1999. Patients will undergo a freeze-all cycle, with no fresh transfer of embryos.

The primary outcome measure will be the total number of mature (MII) oocytes available for cryopreservation.

Secondary outcome measures will include the following:

* Total number of oocytes retrieved per cycle
* Ratio of mature (MII) to immature oocytes
* Total number of mature oocytes (MII) retrieved per IVF/ICSI cycle
* Ratio of mature (MII) to immature oocytes per IVF/ICSI cycle
* Number of two pronuclei (2PN) zygotes
* Fertilization rate, which will include two outcomes each defined as follows:

Definition 1: number of 2PN zygotes divided by the number of mature oocyte(s) fertilized per IVF/ICSI cycle.

Definition 2: number of 2PN zygotes divided by the number of oocytes incubated with at least 10,000 sperm per IVF cycle.

* Total number of day 3 embryos
* Total number of good quality day 5 embryos available for cryopreservation determined by a blinded embryologist using the classification system by Gardner and Schoolcraft, 1999.
* Incidence of moderate to critical OHSS based on the classification criteria by Mathur et al. 2005

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40.
* Undergoing IVF for fertility preservation (freezing all oocytes or embryos)
* Diagnosed with a non-hormone sensitive malignancy (malignancy other than breast, uterine and ovarian cancer)
* GnRH antagonist protocol (standard of care for all fertility preservation patients)

Exclusion Criteria:

* Any contraindication to treatment with gonadotropins (including medical history or risk factors for TE, hypersensitivity to gonadotropins or to any of the excipients).
* Congenital hypogonadotropic hypogonadism unrelated to the oncological condition.
* Previous adverse or allergic reaction to luteinizing hormone or any of its drug components.
* Had prior radiotherapy to the abdomen or pelvis
* Prior chemotherapy
* Prior history of deep vein thrombosis, or pulmonary embolism
* Patients with a diagnosis of hormone sensitive cancer including ovarian, uterine, or mammary carcinoma
* Patients with uncontrolled thyroid or adrenal failure
* Patients with active, untreated tumors of the hypothalamus and pituitary gland
* Patients who are lactating
* Patients with a known diagnosis of primary ovarian failure
* Previous participant of this study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Total number of mature (MII) oocytes available for cryopreservation | 12hrs after egg retrieval

SECONDARY OUTCOMES:
Total number of oocytes retrieved per cycle | 1hr after egg retrieval
Ratio of mature (MII) to immature oocytes | 12 hours after egg retrieval
Total number of mature oocytes (MII) retrieved per IVF/ICSI cycle | 12 hours after egg retrieval
Ratio of mature (MII) to immature oocytes per IVF/ICSI cycle | 12 hours after egg retrieval
Number of two pronuclei (2PN) zygotes | 48 hours after egg retrieval
Fertilization rate, which will include two outcomes each defined as follows: | 48 hours after egg retrieval
  * Definition 1: number of 2PN zygotes divided by the number of mature oocyte(s) fertilized per IVF/ICSI cycle.
  * Definition 2: number of 2PN zygotes divided by the number of oocytes incubated with at least 10,000 sperm per IVF cycle.
Total number of day 3 embryos | 72-80 hours after egg retrieval
Total number of good quality day 5 embryos available for cryopreservation determined by a blinded embryologist using the classification system by Gardner and Schoolcraft, 1999. | 120-132 hours after egg retrieval
Incidence of moderate to critical OHSS based on the classification criteria by Mathur et al. 2005 | 2 weeks after egg retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Greenblatt, MD FRCSC, Principal Investigator — Mount Sinai Fertility, Mount Sinai Hospital, University of Toronto

IPD SHARING:
Plan to Share IPD: Yes
All IPD datasets that underlie results in the publication will be shared, including study protocol, statistical analysis plan, and clinical study plan.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 6 months after article publication and data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
  For more information or to submit a request, please contact swati.dixit@sinaihealth.ca.

DOCUMENTS (1):
  • Study Protocol (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT06227949/Prot_000.pdf